CLINICAL TRIAL: NCT03063450
Title: CheckpOiNt Blockade For Inhibition of Relapsed Mesothelioma (CONFIRM): A Phase III Double-Blind, Placebo Controlled Trial to Evaluate the Efficacy of Nivolumab in Relapsed Mesothelioma
Brief Title: CheckpOiNt Blockade For Inhibition of Relapsed Mesothelioma
Acronym: CONFIRM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Southampton (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22864; 2016-003111-35 (EudraCT Number); CA209-841 (Other Grant/Funding Number: Bristol-Myers Squibb); A21400 (Other Grant/Funding Number: Cancer Research UK)
Record Dates: First submitted 2017-02-10; First posted 2017-02-24 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2024-05

CONDITIONS: Mesothelioma
Keywords: anti PD-L1; nivolumab; immunotherapy; RECIST; quality of life; survival; immune checkpoint inhibition
MeSH Terms: conditions — Mesothelioma | interventions — Nivolumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nivolumab (Experimental): Nivolumab 240mg flat dose Q2W over 30 minutes IV until disease progression, to a maximum of 12 months
  Interventions: Drug: Nivolumab
- Placebo (Placebo Comparator): Sterile 0.9% sodium chloride Q2W over 30 minutes IV until disease progression, to a maximum of 12 months
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Nivolumab — Nivolumab at a dose of 240mg as a 30-minute IV infusion, on Day 1 of every 14 day treatment cycle
  Other Names: Opdivo
  Arms: Nivolumab
Other: Placebo — Placebo consisting of sterile 0.9% sodium chloride as a 30-minute IV infusion, on Day 1 of every 14 day treatment cycle
  Arms: Placebo

SUMMARY:
The UK has the highest incidence of mesothelioma. The incidence has risen by 497% since the late 1970's and is increasing worldwide due to continued mining and use of asbestos. For patients with mesothelioma who have relapsed after taking pemetrexed and cisplatin, there is currently no standard treatment, making this an urgent unmet need. Recent trials in this area have not found an effective treatment that improves overall survival.

Following a debate in the House of Lords, a national survey assessing the research priorities in mesothelioma found that 'exploiting the potential of immunotherapy' was a top priority. This trial was designed in response to that survey. It uses the immunotherapy agent nivolumab which blocks programmed cell death 1 (PD-1) receptor on activated T-cells (a type of white blood cell forming part of the immune system). Early research has found a dependency of mesothelioma on the PD-1 checkpoint. By attaching to PD-1, nivolumab blocks its action (checkpoint inhibition), preventing it from turning off the T-cell, and therefore allowing the immune system to work. PD-1 checkpoint inhibition has revolutionised the treatment of melanoma and it is hoped to be as effective in mesothelioma.

This trial is a randomised, double blind placebo controlled trial of patients with mesothelioma who are second or third relapse following a platinum based chemotherapy treatment.

DETAILED DESCRIPTION:
Effective therapy for relapsed mesothelioma is an unmet need. Despite a significant number of clinical studies in the second line setting, no randomised study to date has been positive. The James Lind Alliance Priority Setting Partnership funded by the NIHR has identified immunotherapy as the number one UK research priority. To date there have been no placebo controlled randomised trials for mesothelioma using PD-L1 or PD-1 checkpoint inhibition. Early promising signals of activity relating to both PD-L1 and PD-1 targeted treatment in mesothelioma implicate a dependency of mesothelioma on this immune checkpoint, and support the development of a randomised phase III trial to evaluate the efficacy of nivolumab. CONFIRM will be the first ever placebo controlled, randomised phase III trial of a PD-1 immune checkpoint inhibitor.

PD-1 checkpoint inhibition has revolutionised the treatment of melanoma and is now standard of care in non-small cell lung cancer, squamous cell cancer head and neck and classical Hodgkin's lymphoma. It is being assessed rigorously in numerous other cancers making its evaluation in mesothelioma timely in CONFIRM.

This trial is a randomised, double blind placebo controlled trial of patients with mesothelioma who are second or third relapse following a platinum based chemotherapy treatment. Patients will be randomised in a 2:1 ratio (nivolumab: placebo).

336 patients will be recruited from 25 UK centres with the last patient having a minimum of 6 months follow up. All patients will be on treatment for 12 months unless they progress or withdrawal prior to this.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated a REC-approved written informed consent form in accordance with regulatory and institutional guidelines. Must be obtained before the performance of any protocol-related procedures that are not part of normal patient care.
* Consent to provide tissue and blood samples for research
* Must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests, and other requirements of the study
* Histological confirmation of mesothelioma (any subtype, pleural or peritoneal).
* Must have received treatment with at least one prior line of treatment. Prior maintenance therapy (e.g. avastin) is allowed and will not count as a line of therapy. Prior lines of antineoplastic therapy, including chemotherapy, surgical resection of lesions, radiation therapy, must be completed within 14 days of receiving nivolumab
* ECOG PS 0-1
* Age ≥18 years
* Expected survival of at least 12 weeks
* Radiologically assessable disease by modified RECIST (pleural mesothelioma) or RECIST 1.1 (non-pleural mesothelioma or where measurements for mRECIST cannot be obtained).
* Evidence of disease progression by CT scan
* Prior palliative radiotherapy must have been completed at least 14 days prior to study drug administration
* Screening laboratory values must meet the following criteria within 48 hours prior to commencement of treatment:

  i) White blood cells ≥ 2 x 10^9/L ii) Neutrophils ≥1.5 x 10^9/L iii) Platelets ≥ 100 X10^9/L iv) Haemoglobin ≥ 90 g/L v) Serum creatinine of ≤ 1.5 X ULN or creatinine clearance (CrCl) > 50 mL/minute (using Cockcroft/Gault formula) vi) AST ≤ 3 X ULN vii) ALT ≤ 3 X ULN viii) Total bilirubin ≤ 1.5 X ULN (except patients with Gilbert Syndrome, who must have total bilirubin < 51.3 μmol/L) 2 x 10^9/L
* Reproductive status

  1. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) at enrolment and within 24 hours prior to the start of study drug.
  2. Women must not be breastfeeding.
  3. WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with nivolumab plus 5 half-lives of nivolumab (5 x half-life=125 days) plus 30 days (duration of ovulatory cycle) for a total of 5 months post- treatment completion.
  4. Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 7 months after the last dose of investigational product. Women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile as well as azoospermic men do not require contraception.
* Expected survival of at least 12 weeks.

Exclusion Criteria:

* Target Disease Exceptions

  1. Patients with untreated, symptomatic CNS metastases are excluded. Participants are eligible if CNS metastases are adequately treated and participants are neurologically returned to baseline (except for residual signs or symptoms related to the CNS treatment) for at least 2 weeks prior to treatment assignment. In addition, participants must be either off corticosteroids, or on a stable or decreasing dose of <=10 mg daily prednisone (or equivalent) for at least 2 weeks prior to treatment.
  2. Patients with carcinomatous meningitis are excluded.
* Physical and Laboratory Test Findings

  1. Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
  2. Any positive test for hepatitis B virus or hepatitis C virus indicating acute or chronic infection.
* Allergies and Adverse Drug Reactions

  a) History of severe hypersensitivity reactions to other monoclonal antibodies
* Medical History and Concurrent Diseases

  1. Patients with active, known or suspected autoimmune disease.
  2. Patients with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of the first dose of study drug administration. Inhaled or topical steroids and adrenal replacement steroid doses > 10 mg daily prednisone or equivalent are permitted in the absence of active autoimmune disease.
  3. Other active malignancy requiring concurrent intervention.
  4. Patients with previous malignancies (except non-melanoma skin cancers, and the following in situ cancers: bladder, gastric, colon, endometrial, cervical/dysplasia, melanoma or breast) are excluded unless a complete remission was achieved at least 2 years prior to study entry AND no additional therapy is required during the study period.
  5. Any serious or uncontrolled medical disorder or active infection that, in the opinion of the investigator, may increase the risk associated with study participation, study drug administration, or would impair the ability of the patient to receive protocol therapy.
  6. All toxicities attributed to prior anti-cancer therapy other than alopecia and fatigue not resolved to Grade 1 (NCI CTCAE version 4.03) or baseline before administration of study drug.
  7. Patients who have not recovered from the effects of major surgery or significant traumatic injury at least 14 days before the first dose of study treatment.
  8. Known alcohol or drug abuse.
  9. Patients who have received prior therapy with anti-PD-1, anti-PD-L1, anti-PD-L2, anti- CD137, or anti-CTLA-4 antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways) or who have previously taken part in a randomised Bristol Myers Squibb (BMS) clinical trial for nivolumab or ipilimumab including study CA209-743 (CheckMate 172) or in the CCTG trial of pembrolizumab (IND.227).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2023-02-07 (Actual); Study Completion 2023-02-07 (Actual)

PRIMARY OUTCOMES:
Overall survival | Time from randomisation to date of death from any cause or time of censoring
  Length of time participants are alive
Progression free survival | Time from randomisation to investigator-reported progression, death, or end of study (max. 12 months from last participant randomised)
  Length of time participants are free of disease progression

SECONDARY OUTCOMES:
Overall response rate (modified RECIST or RECIST 1.1) | From randomisation and while on treatment
  Response of disease to treatment
EQ-5D-5L | At baseline, after cycles 3 and 6 (each cycle is 14 days) and 1, 6 and 12 months post progression/treatment discontinuation.
  Quality of life
CTCAE V4.03 | At baseline, after each treatment cycle (each cycle is 14 days) and each follow up visit. Up to 30 days post progression/treatment discontinuation.
  Adverse events
Health resource use | Up to max. 24 months. At baseline, after cycles 3 and 6 (each cycle is 14 days) and 1, 6 and 12 months post progression/treatment discontinuation.
  Bespoke health resource use questionnaire capturing information on hospital visits.
Progression-free survival (RECIST) | From randomisation until 28 days after completing treatment (max. 12 months), progression, or death
  Time participant is free of disease progression, as measured by RECIST

OTHER OUTCOMES:
Translational | Samples collected at baseline and optional sample at progression (assessed up to 51 months from randomisation)
  To correlate:
  1. mutation burden with OS
  2. immunosuppressive landscape (immune checkpoint expression and infiltration of immune cell) and nivolumab efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Dean Fennell, Principal Investigator — University of Leicester; Gareth Griffiths, Principal Investigator — Southampton Clinical Trials Unit, University of Southampton
Locations (24):
- United Kingdom (24):
  - Ulster Hospital, Dundonald, Belfast
  - Raigmore Hospital, Inverness, Inverness
  - East Kent Hospitals University Foundation Trust, Canterbury, Kent
  - Northumbria Healthcare NHS Foundation Trust, Newcastle upon Tyne, Northumberland
  - Aberdeen Royal Infirmary, Aberdeen
  - Basildon University Hospital, Basildon
  - Belfast City Hospital, Belfast
  - Royal Bournemouth Hospital, Bournemouth
  - Addenbrooke's Hospital, Cambridge
  - Velindre Cancer Centre, Cardiff
  - Ninewells Hospital, Dundee
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Harrogate District Hospital, Harrogate
  - University Hospitals Morecambe Bay, Lancaster
  - Leicester Royal Infirmary, Leicester
  - Barts Cancer Institute, London
  - University College London Hospitals NHS Foundation Trust, London
  - Wythenshawe Hospital, Manchester
  - Mount Vernon Cancer Centre, Northwood
  - Churchill Hopsital, Oxford
  - Southampton General Hospital, Southampton
  - Southend Hospital, Southend-on-Sea
  - Lister Hospital, Stevenage
  - Musgrove Park Hospital, Taunton

IPD SHARING:
Plan to Share IPD: Yes
As a minimum, anonymous data will be available for request from three months after publication of an article, to researchers who provide a completed Data Sharing request form that describes a methodologically sound proposal, for the purpose of the approved proposal and if appropriate a signed Data Sharing Agreement. Data will be shared once all parties have signed relevant data sharing documentation.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be shared once all parties have signed relevant data sharing documentation, from three months following publication of the final analysis.
Access Criteria: Completion of data access request via Southampton CTU website.
URL: http://www.southampton.ac.uk/ctu

REFERENCES:
- [Background] Fennell DA, Kirkpatrick E, Cozens K, Nye M, Lester J, Hanna G, Steele N, Szlosarek P, Danson S, Lord J, Ottensmeier C, Barnes D, Hill S, Kalevras M, Maishman T, Griffiths G. CONFIRM: a double-blind, placebo-controlled phase III clinical trial investigating the effect of nivolumab in patients with relapsed mesothelioma: study protocol for a randomised controlled trial. Trials. 2018 Apr 18;19(1):233. doi: 10.1186/s13063-018-2602-y. PMID 29669604
- [Derived] Fennell DA, Ewings S, Ottensmeier C, Califano R, Hanna GG, Hill K, Danson S, Steele N, Nye M, Johnson L, Lord J, Middleton C, Szlosarek P, Chan S, Gaba A, Darlison L, Wells-Jordan P, Richards C, Poile C, Lester JF, Griffiths G; CONFIRM trial investigators. Nivolumab versus placebo in patients with relapsed malignant mesothelioma (CONFIRM): a multicentre, double-blind, randomised, phase 3 trial. Lancet Oncol. 2021 Nov;22(11):1530-1540. doi: 10.1016/S1470-2045(21)00471-X. Epub 2021 Oct 14. PMID 34656227
- See also: Preliminary data for the trial — https://doi.org/10.1016/S1470-2045(21)00471-X